CLINICAL TRIAL: NCT03111914
Title: Applications of Dual Energy CT for Improving Staging and Monitoring of Therapy Response in Patients With Osseous Metastases From Castrate-resistant Prostate Cancer
Brief Title: Applications of Dual Energy CT in Patients With Osseous Metastases From Castrate-resistant Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary Issues
Sponsor: Duke University (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00078046
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Dual Energy CT (DECT); Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dual Energy Computed Tomography (DECT) (Other): This is a single-arm study. Each patient will receive an unenhanced dual energy CT scan followed by a contrast-enhanced scan as part of clinical routine work up. No change in the contrast material injection protocol will be performed for this this study.
  Interventions: Diagnostic Test: Dual Energy Computed Tomography

INTERVENTIONS:
Diagnostic Test: Dual Energy Computed Tomography — The subject's diagnostic scan will be preceded by a not clinically indicated non enhanced dual energy scan. The overall radiation dose to the patient for the first and second acquisition will be twice the radiation dose of a conventional CT of the chest, abdomen and pelvis. The non enhanced dual energy scan will be repeated during a clinical follow-up after the subject's first three months of enrollment and at a clinical follow-up after six months of enrollment.
  The clinically-indicated, contrast-enhanced diagnostic scan will be performed according to standard of care.
  Other Names: DECT

SUMMARY:
The purpose of this study is to establish a more accurate and precise way to image (take pictures of) metastatic bone disease in patients with prostate cancer for staging and monitoring response to therapy. More specifically, the study aims to evaluate the capabilities of dual energy CT as a more precise and accurate tool for staging and monitoring of therapy response in patients with osseous metastases from castrate-resistant prostate cancer.

Bone metastases in prostate cancer patients are a clinical and diagnostic challenge to image. Sometimes very small metastatic bone lesions may only become detectable by imaging in response to therapy due to increased bone deposition during the first three months after therapy. Commonly used imaging tests (such as regular CT or bone scan) are unable to reliably tell the difference between increased bone deposition (therapy response) and growth of the lesion (progressive disease). This diagnostic challenge may have profound negative effects on patient management since it may require additional imaging before an accurate determination of tumor response can be made. An appropriate determination of tumor response is needed for appropriate management of prostate cancer. The investigators anticipate that the new imaging tested in this study (called dual energy CT) may provide additional critical information in this clinical and diagnostic challenge.

Approximately 100 people with prostate cancer and metastatic bone disease will take part in this study. At enrollment, three months, and six months, they will will receive a non-enhanced (without contrast) dual energy CT scan of the chest, abdomen and pelvis before receiving their routine, clinical contrast-enhanced CT scan.

ELIGIBILITY:
Inclusion Criteria:

1. Oncology patients with castrate-resistant prostate cancer planned for therapy with abiraterone acetate or enzalutamide and prednisolone undergoing clinically indicated MDCT (multi-detector computed tomography) of the chest, abdomen and pelvis
2. > 18 years old
3. Serum creatinine < 2.0
4. BMI < 35kg/m^2
5. Sign informed consent

Exclusion Criteria:

- History of anaphylactoid reaction to iodinated contrast material

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dual Energy Computed Tomography (DECT): This is a single-arm study. Each patient will receive an unenhanced dual energy CT scan followed by a contrast-enhanced scan as part of clinical routine work up. No change in the contrast material injection protocol will be performed for this this study.
  Dual Energy Computed Tomography: The subject's diagnostic scan will be preceded by a not clinically indicated non enhanced dual energy scan. The overall radiation dose to the patient for the first and second acquisition will be twice the radiation dose of a conventional CT of the chest, abdomen and pelvis. The non enhanced dual energy scan will be repeated during a clinical follow-up after the subject's first three months of enrollment and at a clinical follow-up after six months of enrollment.
  The clinically-indicated, contrast-enhanced diagnostic scan will be performed according to standard of care.
Period: Overall Study
Arm/Group | Dual Energy Computed Tomography (DECT)
Started | 7
Completed | 0
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Due to the complexity and challenges in spatial resolution of clinical CT images, the intended analysis failed to differentiate between normal and abnormal bone marrow changes which precluded an accurate analysis of treatment effects. A consensus decision was made to stop recruitment until technical challenges have been solved.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Optimal Threshold for Iodine Uptake to Differentiate Between Therapy Response and Progression of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

2. Primary Outcome: Sensitivity of Optimal Threshold for Iodine Uptake to Differentiate Between Therapy Response and Progression of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

3. Primary Outcome: Specificity of Optimal Threshold for Iodine Uptake to Differentiate Between Therapy Response and Progression of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

4. Primary Outcome: Accuracy of Optimal Threshold for Iodine Uptake to Differentiate Between Therapy Response and Progression of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

5. Primary Outcome: Reader Performance for Iodine Maps and Fused Images to Differentiate Between Therapy Response and Progression of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

6. Primary Outcome: Sensitivity of Imaging Approach
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

7. Primary Outcome: Specificity of Imaging Approach
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

8. Primary Outcome: Accuracy of Imaging Approach
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

9. Secondary Outcome: Optimal Threshold for Iodine Uptake to Diagnose of Metastatic Bone Disease.
Description: To analyze the feasibility to detect bone metastasis at baseline more accurately, unenhanced bone marrow imaging will be calculated and additional dual energy based, calcium corrected iodine maps will be used to determine a threshold for detection of vital bone metastasis in order to calculate color coded bone maps for risk of presence of bone metastases.
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

10. Secondary Outcome: Reader Performance for Iodine Maps and Fused Images to Diagnose Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

11. Secondary Outcome: Sensitivity of Optimal Threshold for Iodine Uptake to Diagnose of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

12. Secondary Outcome: Specificity of Optimal Threshold for Iodine Uptake to Diagnose of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

13. Secondary Outcome: Accuracy of Optimal Threshold for Iodine Uptake to Diagnose of Metastatic Bone Disease
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

14. Secondary Outcome: Optimal Threshold for Iodine Uptake to Diagnose Metastatic Lymph Nodes
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

15. Secondary Outcome: Sensitivity of Optimal Threshold for Iodine Uptake to Diagnose Metastatic Lymph Nodes
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

16. Secondary Outcome: Specificity of Optimal Threshold for Iodine Uptake to Diagnose Metastatic Lymph Nodes
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

17. Secondary Outcome: Accuracy of Optimal Threshold for Iodine Uptake to Diagnose Metastatic Lymph Nodes
Description: Feasibility of monitoring metastatic bone disease in prostate cancer patients
Time Frame: Duration of CT scan (approximately 5 minutes)
Population: Data not collected due to technical issues.
Arm/Group | Dual Energy Computed Tomography (DECT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | Dual Energy Computed Tomography (DECT)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Due to the complexity and challenges in spatial resolution of clinical CT images, the intended analysis failed to differentiate between normal and abnormal bone marrow changes which precluded an accurate analysis of treatment effects. A consensus decision was made to stop recruitment until technical challenges have been solved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03111914/Prot_SAP_000.pdf